CLINICAL TRIAL: NCT00339573
Title: National Survey of Lead Hazards and Allergens in Housing
Brief Title: National Survey of Lead and Allergen Hazards in Housing
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998033; OH98-E-N033
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Asthma; Allergy
Keywords: Asthma; Exposure; Home; Indoor; Allergy
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- National Housing Stock: The target population of this study was the national housing stock (1998-1999) ofapproximately 95 million housing units.

SUMMARY:
We propose to conduct a scientifically valid, descriptive survey to measure the prevalence and levels of lead in dust, soil, and paint, and the prevalence and levels of various indoor allergens in floor and bedding dust in the nation's housing stock. The survey strategy is a population-based, multi-stage area probability sample designed to represent all 50 states. The survey will include approximately 1000 homes in at least 100 primary sampling units (PSU, a metropolitan area or cluster of counties). Residents of candidate participant housing units (HUs) will initially be contacted by a letter to introduce and provide a brief explanation of the study. A field interviewer will then visit each candidate HU to screen and recruit eligible units into the study. A short Screening Questionnaire will be administered to an adult HU resident and an invitation will be extended to those HUs that are eligible to participate in the study. A field data collection visit will be scheduled for the following week, at the resident's convenience. The collection visit will be conducted by two member team (including the same field interviewer that will conduct the screening/recruiting visit) and will consist of administration of an informed consent form and Data Collection Questionnaire, completion of home observation forms, collection of interior dust and exterior soil samples, and conduct of nondestructive paint lead analysis on both interior and exterior walls. Soil and dust samples will be shipped to analytical laboratories for lead and allergen analysis. Extensive survey design, procedure, and reporting details are provided in the National Survey Lead Hazards and Allergens in Housing: Protocol and Sample Design Report (Attachment A). It is anticipated that this study will provide allergen-specific data regarding: 1) housing conditions, demographic factors, and climate to facilitate evaluation of regional, ethnic, socioeconomic, and housing characteristic differences in the indoor allergen burden; 2) an estimate of indoor allergen exposure in the U.S. population; 3) baseline data that can be used to stimulate future studies which attempt to correlate allergen exposure to disease outcome. The study will yield lead hazard data to: 1) estimate the number and percent of homes with dust and soil lead levels above selected thresholds; 2) identify sources of lead in dust in housing; 3) permit future analysis of lead hazard control strategies an costs, including associated policy and regulatory guidelines.

DETAILED DESCRIPTION:
We propose to conduct a scientifically valid, descriptive survey to measure the prevalence and levels of lead in dust, soil, and paint, and the prevalence and levels of various indoor allergens in floor and bedding dust in the nation's housing stock. The survey strategy is a population-based, multi-stage area probability sample designed to represent all 50 states. The survey will include approximately 1000 homes in at least 100 primary sampling units (PSU, a metropolitan area or cluster of counties). Residents of candidate participant housing units (HUs) will initially be contacted by a letter to introduce and provide a brief explanation of the study. A field interviewer will then visit each candidate HU to screen and recruit eligible units into the study. A short Screening Questionnaire will be administered to an adult HU resident and an invitation will be extended to those HUs that are eligible to participate in the study. A field data collection visit will be scheduled for the following week, at the resident's convenience. The collection visit will be conducted by a two member team (including the same field interviewer that will conduct the screening/recruiting visit) and will consist of administration of an informed consent form and Data Collection Questionnaire, completion of home observation forms, collection of interior dust and exterior soil samples, and conduct of nondestructive paint lead analyses on both interior and exterior walls. Soil and dust samples will be shipped to analytical laboratories for lead and allergen analysis. Extensive survey design, procedure, and reporting details are provided in the National Survey Lead Hazards and Allergens in Housing: Protocol and Sample Design Report. It is anticipated that this study will provide allergen-specific data regarding: 1) housing conditions, demographic factors, and climate to facilitate evaluation of regional, ethnic, socioeconomic, and housing characteristic differences in the indoor allergen burden; 2) an estimate of indoor allergen exposure in the U.S. population; 3) baseline data that can be used as a reference point for future allergen surveys; and 4) a database that can be used to stimulate future studies which attempt to correlate allergen exposure to disease outcome. The study will yield lead hazard data to: 1) estimate the number and percent of homes with dust and soil lead levels above selected thresholds; 2) identify sources of lead in dust in housing; 3) permit future analysis of lead hazard control strategies and costs, including associated policy and regulatory guidelines.

ELIGIBILITY:
* INCLUSION CRITERIA:

The target population for the Survey is the national housing stock of approximately 95 million housing units.

The decision to include or exclude a subset is usually based on such factors as relevancy to the study objectives, availability of data from other sources, and effort required to obtain the study data.

None of the possible housing type exclusion or oversampling proposals are based upon gender, race, ethnic, cultural, or biological factors.

Housing built after 1977.

Housing units in multi-family buildings.

Manufactured housing units, i.e., mobile homes and trailers.

EXCLUSION CRITERIA:

Housing where children are not permitted to live (elderly housing, nursing homes, college dormitories, etc.).

Group housing - both institutional (prisons or jails, detention centers, hospitals, military housing, etc.) and non-institutional (dormitories, fraternities, orphanages, rooming houses, missions, work camps, convents, etc.).

Vacant housing.

Short-term housing. This category includes homes which are not the resident's sole or permanent home, and which the resident present at the time of field data collection spends less than three months per year. This includes seasonal, occasional use, recreational, and second homes, as well as homes for migrant workers.

Hotels and motels.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A nationally representative sample of 831 housing units, inhabited by 2,456 individuals, within 75 different locations throughout the US was surveyed.
Sampling Method: Probability Sample
Enrollment: 831 (Actual)
Dates: Start 1998-06-30 (Actual); Primary Completion 1999-08-31 (Actual); Study Completion 1999-08-31 (Actual)

PRIMARY OUTCOMES:
Concentrations of indoor allergens and lead | Cross-sectional assessment during the field visit
  The primary outcomes included concentrations of common indoor allergens (dust mite, cat, dog, cockroach, mouse, and Alternaria) in household dust and lead levels in paint, household dust, and soil in the nation's housing.

CONTACTS AND LOCATIONS:
Overall Officials: Darryl C Zeldin, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Needleman HL, Gatsonis CA. Low-level lead exposure and the IQ of children. A meta-analysis of modern studies. JAMA. 1990 Feb 2;263(5):673-8. PMID 2136923
- [Background] Pocock SJ, Smith M, Baghurst P. Environmental lead and children's intelligence: a systematic review of the epidemiological evidence. BMJ. 1994 Nov 5;309(6963):1189-97. doi: 10.1136/bmj.309.6963.1189. PMID 7987149
- [Background] Pollart SM, Mullins DE, Vailes LD, Hayden ML, Platts-Mills TA, Sutherland WM, Chapman MD. Identification, quantitation, and purification of cockroach allergens using monoclonal antibodies. J Allergy Clin Immunol. 1991 Feb;87(2):511-21. doi: 10.1016/0091-6749(91)90010-l. PMID 1993811